CLINICAL TRIAL: NCT04974489
Title: Correcting Public Misperceptions About Very Low Nicotine Content Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-1284; R21CA234968 (NIH)
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Tobacco Use, Cigarette Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Emotion-based messages about the harm of VLNC (Experimental)
  Interventions: Behavioral: Emotion-based messages about the harm of VLNC
- Continued-harm-framed messages about the harm of VLNC (Experimental)
  Interventions: Behavioral: Continued-harm-framed messages about the harm of VLNC
- Myth-refuting messages about the harm of VLNC (Experimental)
  Interventions: Behavioral: Myth-refuting messages about the harm of VLNC
- Control messages about littering (Active Comparator)
  Interventions: Behavioral: Control messages about littering

INTERVENTIONS:
Behavioral: Emotion-based messages about the harm of VLNC — Participants in this arm will receive 3 emotion-based messages about the harm of VLNC during the survey data collection.
  Arms: Emotion-based messages about the harm of VLNC
Behavioral: Continued-harm-framed messages about the harm of VLNC — Participants in this arm will receive 3 continued-harm-framed messages about the harm of VLNC during the survey data collection.
  Arms: Continued-harm-framed messages about the harm of VLNC
Behavioral: Myth-refuting messages about the harm of VLNC — Participants in this arm will receive 3 myth-refuting messages messages about the harm of VLNC during the survey data collection.
  Arms: Myth-refuting messages about the harm of VLNC
Behavioral: Control messages about littering — Participants in this arm will receive 3 control messages about littering during the survey data collection.
  Arms: Control messages about littering

SUMMARY:
Tobacco use is the leading preventable cause of cancer and cancer deaths in the US. While most (69%) smokers want to quit, only 6% succeed in doing so each year. For many smokers, the addictiveness of nicotine makes quitting very difficult. To reduce cigarette smoking and resulting harms, FDA has announced a comprehensive approach to tobacco and nicotine regulation that includes moving toward a very low nicotine content (VLNC) standard for cigarettes. Greatly reduced nicotine levels would facilitate smoking cessation. However, the maximal success of the policy may require public understanding that, although these new cigarettes are less addictive, their high toxicity and carcinogenicity are unchanged. Yet, nearly half of adult smokers incorrectly think smoking VLNC cigarettes is less harmful than smoking current cigarettes (the VLNC misperception). Additionally, 24% of smokers said they would be less likely to quit if a VLNC regulation is enacted. Thus, the VLNC misperception may partially undermine a nicotine reduction policy. Although communication research suggests it is challenging to change people's incorrect understanding, new communication techniques may help reduce the VLNC misperception. In this randomized trial we will examine whether messages about the harm of VLNC cigarettes can reduce the VLNC misperception and increase intention to quit in a nicotine reduction scenario.

DETAILED DESCRIPTION:
In this study we will assess whether messages about the harm of VLNC cigarettes reduce the misperception that they are less harmful than regular cigarettes.

Recruitment:

We will enroll participants from an existing nationally representative panel.

Informed Consent:

Potential participants are part of an existing nationally representative panel and have already consented to participate in the panel. Before enrolling, participants will also be asked to consent to participate in this study via a consent form included in the study survey.

Randomization:

Survey software will randomly allocate participants to one of the four arms of the study (3 intervention arms or a control arm). Each study arm will have approximately the same number of participants.

Assessment:

Participants will complete a 15-minute survey. The survey will begin with an introduction to the concept of VLNC cigarettes. Then participants will be shown intervention or control messages, and their beliefs will be assessed.

Detailed Description of the Intervention:

Participants will be shown a set of 3 messages about the harms of VLNC cigarettes (intervention arms) or about littering (control arm). Each of the 3 intervention arms use a different theme to attempt to correct the VLNC misperception.

ELIGIBILITY:
Inclusion Criteria:

* Current Cigarette Smoker
* Age 18 or older
* Enrolled in existing nationally representative panel where recruitment is based

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1153 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Justin Byron, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a panel, screened for study eligibility, and invited to enroll after they were determined to be eligible.
Pre-assignment Details: 1,253 participants completed the study questionnaire, and the panel provider determined that of those 1,145 qualified participants completed the questionnaire. The panel provider removed 13 cases from the study who skipped half or more of the survey questions. The study team received data for 1,132 participants. For analysis purposes, we excluded anyone who did not complete the questions for the primary outcome (n=79), yielding a final analysis sample size of 1,053.
Period: Overall Study
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Started (Participants included in the sample sent from the panel provider to the study team.) | 285 | 274 | 288 | 285
Completed | 262 | 261 | 263 | 267
Not Completed | 23 | 13 | 25 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering | Total
Number analyzed (Participants) | 262 | 261 | 263 | 267 | 1053
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (13.7) | 54.6 (13.6) | 54.4 (13.2) | 54.9 (13.1) | 54.5 (13.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 138 | 131 | 129 | 136 | 534
  Female | 122 | 129 | 134 | 127 | 512
  Non-binary and Prefer to Self Describe | 1 | 0 | 0 | 4 | 5
  Missing | 1 | 1 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 201 | 203 | 192 | 197 | 793
  Black, Non-Hispanic | 22 | 27 | 39 | 35 | 123
  Hispanic or Latino | 22 | 19 | 23 | 19 | 83
  Other, Non-Hispanic | 9 | 4 | 4 | 6 | 23
  Two Races or More, Non-Hispanic | 8 | 8 | 5 | 10 | 31
Region of Enrollment [Number; unit: participants]
  United States | 262 | 261 | 263 | 267 | 1053

OUTCOME MEASURES:

1. Primary Outcome: Very Low Nicotine Content (VLNC) Misperception
Description: Measured by a 3 item scale. Very low nicotine content (VLNC) Misperception measured with 3 questions, the final VLNC misperception score is a mean of the response to the 3 questions, on a scale of 1 to 5, where 1 indicates a perception that VLNC are much more harmful than other cigarettes, and 5 indicates a perception that VLNC are much less harmful than other cigarettes, and 3 is a perception that VLNC are as harmful as other cigarettes.
Time Frame: During one day survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 262 | 261 | 263 | 267
score on a scale | 3.12 (0.56) | 3.04 (0.61) | 3.04 (0.54) | 3.36 (0.80)

2. Secondary Outcome: Quit Intentions
Description: Measured by a 3 item scale. Quit intention measured with 3 questions, the final quit intention score is a mean of the response to the 3 questions, on a scale of 1 to 5, where 1 indicates low intention to quit smoking, and 5 indicates a high intention to quit.
Time Frame: During one day survey
Population: Overall number of participants analyzed is the number of participants in each condition that responded to all 3 questions for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 255 | 251 | 258 | 258
score on a scale | 2.88 (1.22) | 2.80 (1.13) | 2.87 (1.27) | 2.85 (1.26)

3. Other Pre Specified Outcome: Perceived Message Effectiveness
Description: Measured by a 3 item scale after each message, 9 items total. Perceived message effectiveness measured with 3 questions per message. The final perceived message effectiveness score is a mean of the response to the 3 questions, on a scale of 1 to 5, where 1 indicates low perceived message effectiveness, and 5 indicates high perceived message effectiveness.
Time Frame: During one day survey
Population: Overall number of participants analyzed is the number of participants in each condition that responded to all 9 questions for the outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 254 | 257 | 257 | 263
score on a scale | 3.07 (0.87) | 3.26 (0.86) | 3.17 (0.90) | 2.45 (0.96)

4. Other Pre Specified Outcome: Perceived Understandability
Description: Perceived Understandability is measured with 1 question on a scale of 1 to 5: "How easy was it to understand the three black and white messages we showed you earlier?", where 1 = "Not at all", 5 = "Very", and 3 = "Somewhat"
Time Frame: During one day survey
Population: Overall number of participants analyzed is the number of participants in each condition that responded to the outcome measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 262 | 261 | 263 | 265
units on a scale | 4.48 (0.82) | 4.5 (0.83) | 4.37 (0.86) | 4.35 (0.94)

5. Other Pre Specified Outcome: Attention
Description: Attention is measured with 1 question on a scale of 1 to 5: "How much did the messages grab your attention?", where 1 = "Not at all", 5 = "Very much", and 3 = "Somewhat"
Time Frame: During one day survey
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 261 | 262 | 261 | 267
units on a scale | 3.26 (1.22) | 2.14 (1.10) | 3.13 (1.16) | 2.73 (1.12)

6. Other Pre Specified Outcome: Negative Affect
Description: Negative affect is measured with 1 question on a scale of 1 to 5: "How much did the messages make you feel scared?", where 1 = "Not at all", 5 = "Very much", and 3 = "Somewhat"
Time Frame: During one day survey
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 262 | 261 | 262 | 266
units on a scale | 2.18 (1.31) | 1.97 (1.15) | 1.93 (1.13) | 1.42 (0.78)

7. Other Pre Specified Outcome: Cognitive Reactions
Description: Cognitive Reactions are measured with 1 question on a scale of 1 to 5: "How much did the messages make you think about the risk of smoking cigarettes that have 95% less nicotine?", where 1 = "Not at all", 5 = "Very much", and 3 = "Somewhat"
Time Frame: During one day survey
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 262 | 260 | 263 | 267
units on a scale | 2.68 (1.29) | 2.68 (1.28) | 2.66 (1.23) | 1.97 (1.11)

8. Other Pre Specified Outcome: Social Interactions
Description: Social Interactions are measured with 1 question on a scale of 1 to 5: "How much would you talk with other people about the messages?", where 1 = "Not at all", 5 = "Very much", and 3 = "Somewhat"
Time Frame: During one day survey
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 262 | 260 | 262 | 267
units on a scale | 2.28 (1.28) | 2.16 (1.16) | 2.24 (1.17) | 2.09 (1.17)

9. Other Pre Specified Outcome: Reactance
Description: Reactance is measured with 1 question on a scale of 1 to 5: "How much do you feel that the messages are trying to manipulate you?", where 1 = "Not at all", 5 = "Very much", and 3 = "Somewhat"
Time Frame: During one day survey
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 262 | 259 | 263 | 266
units on a scale | 2.81 (1.41) | 2.61 (1.40) | 2.62 (1.36) | 2.44 (1.33)

10. Other Pre Specified Outcome: Interest in Other Nicotine Products
Description: Measured by a 3 item scale. Interest in other nicotine products with 3 questions, the final score is a mean of the response to the 3 questions, on a scale of 1 to 5, where 1 indicates low interest in other nicotine products, and 5 indicates a high interest in other nicotine products.
Time Frame: During one day survey
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 259 | 258 | 262 | 266
score on a scale | 2.75 (0.86) | 2.80 (0.78) | 2.77 (0.85) | 2.66 (0.84)

11. Primary Outcome: Percentage of Participants With Very Low Nicotine Content (VLNC) Misperception About Harm (Dichotomized)
Description: Very low nicotine content (VLNC) Misperception of Harm was measured with 1 question, on a scale of 1 to 5, where 1 indicates a perception that VLNC are much more harmful than other cigarettes, and 5 indicates a perception that VLNC are much less harmful than other cigarettes, and 3 is a perception that VLNC are as harmful as other cigarettes. The results were dichotomized to indicate the percentage of people who hold the misperception. Specifically, responses of "much less likely" (5) or "less likely" (4) were recoded as 1 (having the misperception), and responses of "Much more likely" (1), "More likely" (2), or "As likely" (3) were recoded as 0 (not having the misperception).
Time Frame: During one day survey
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 262 | 261 | 263 | 267
percentage of participants | 18.3 [13.6 to 23.0] | 12.6 [8.6 to 16.7] | 11.4 [7.5 to 15.3] | 38.2 [32.3 to 44.1]

12. Primary Outcome: Percentage of Participants With Very Low Nicotine Content (VLNC) Misperception About Cancer (Dichotomized)
Description: Very low nicotine content (VLNC) Misperception of Risk of Cancer was measured with 1 question, on a scale of 1 to 5, where 1 indicates a perception that VLNC are much more likely to cause cancer than other cigarettes, and 5 indicates a perception that VLNC are much less likely to cause cancer than other cigarettes, and 3 is a perception that VLNC are as likely to cause cancer as other cigarettes. The results were dichotomized to indicate the percentage of people who hold the misperception. Specifically, responses of "much less likely" (5) or "less likely" (4) were recoded as 1 (having the misperception), and responses of "Much more likely" (1), "More likely" (2), or "As likely" (3) were recoded as 0 (not having the misperception).
Time Frame: During one day survey
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 262 | 261 | 263 | 267
percentage of participants | 16.8 [12.2 to 21.4] | 11.1 [7.3 to 14.9] | 9.5 [5.9 to 13.1] | 31.8 [26.2 to 37.5]

13. Primary Outcome: Percentage of Participants With Very Low Nicotine Content (VLNC) Misperception About Death (Dichotomized)
Description: Very low nicotine content (VLNC) Misperception of Risk of Death was measured with 1 question, on a scale of 1 to 5, where 1 indicates a perception that VLNC are much more likely to cause death than other cigarettes, and 5 indicates a perception that VLNC are much less likely to cause death than other cigarettes, and 3 is a perception that VLNC are as likely to cause death as other cigarettes. The results were dichotomized to indicate the percentage of people who hold the misperception. Specifically, responses of "much less likely" (5) or "less likely" (4) were recoded as 1 (having the misperception), and responses of "Much more likely" (1), "More likely" (2), or "As likely" (3) were recoded as 0 (not having the misperception).
Time Frame: During one day survey
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
Number analyzed (Participants) | 262 | 261 | 263 | 267
percentage of participants | 16.4 [11.9 to 20.9] | 16.1 [11.6 to 20.6] | 9.9 [6.3 to 13.5] | 34.5 [28.7 to 40.2]

ADVERSE EVENTS:
Time Frame: Low risk study, no adverse event data collected
Description: Low risk study, no adverse event data collected
Arm/Group | Emotion-based Messages About the Harm of VLNC | Continued-harm-framed Messages About the Harm of VLNC | Myth-refuting Messages About the Harm of VLNC | Control Messages About Littering
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT04974489/Prot_SAP_000.pdf